CLINICAL TRIAL: NCT03525236
Title: Product Validation by Cancer Patients - Oncoflavour
Brief Title: The Oncoflavour Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Nutricia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201700363
Record Dates: First submitted 2018-04-26; First posted 2018-05-15 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taste of 5 flavors (Experimental): * Each patient will taste 5 products, in sequential-monadic test, randomized, one by one.
  * Patients will take few sips of each study product, ideally in isolation (avoid influence of other patients)
  * For each product tasted the subjects will be asked to answer a questionnaire including 1 question on the palatability of the product using a 10-point hedonic scale and a more detailed organoleptic evaluation of the product.
  * Between product tastings, participants will have a 10 minutes break to rinse their mouth and fill in a questionnaire assessing sensory changes
  Interventions: Other: Tasting of flavours

INTERVENTIONS:
Other: Tasting of flavours — * Each patient will taste 5 products, in sequential-monadic test, randomized, one by one.
  * Patients will take few sips of each study product, ideally in isolation (avoid influence of other patients)
  * For each product tasted the subjects will be asked to answer a questionnaire including 1 question on the palatability of the product using a 10-point hedonic scale and a more detailed organoleptic evaluation of the product.
  * Between product tastings, participants will have a 10 minutes break to rinse their mouth and fill in a questionnaire assessing sensory changes

SUMMARY:
Oral nutritional supplements (ONS) are often prescribed for malnourished patients to help improve nutritional status. Commonly in cancer patients taste and smell alterations and side effects of treatment can affect the palatability and compliance to ONS. A variety of flavours and styles are available of ONS however research of the palatability of these in cancer patients is limited. This study aims to evaluate specific flavours created based on the taste changes occuring during treatment.

We aim to evaluate the patient liking and evaluation of 5 flavors in 3 different types of flavour-sensations:

* Warming/spicy sensation: to trigger the senses and bring new sensations
* Cooling/fresh sensation: to have a fresh mouthfeel and lighter base perception
* Neutral: to avoid that patients experience additional flavour and let them the opportunity to mix it with other food

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Ability to complete and comprehend questionnaires provided
* Undergoing systemic cancer treatment (chemotherapy or concurrent chemoradiotherapy, radiotherapy, targeted therapy or immunotherapy)

Exclusion Criteria:

* Uncertainty about the willingness or ability of the patient to comply with the protocol requirements (no impairment and no cognitive impairments)
* Coexisting-morbidities affecting taste or smell function
* Lactose Intolerance or Galactosaemia
* Dysphagia
* Diabetics
* Food allergies/intolerances to ingredients present in the product
* No rejection of lemon, red fruits, exotic fruit, yellow fruit flavours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Liking of 5 different oral nutritional supplements with adapted flavors | 20 minutes
  To evaluate patient liking and perception about 5 new flavors on a 10-point scale via a sip test

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, Prof, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Haan JJ, Renken RJ, Moshage Y, Kluifhooft DA, Corbier C, Daly LE, Blanchard H, Reyners AKL. Self-reported taste and smell alterations and the liking of oral nutritional supplements with sensory-adapted flavors in cancer patients receiving systemic antitumor treatment. Support Care Cancer. 2021 Oct;29(10):5691-5699. doi: 10.1007/s00520-021-06049-4. Epub 2021 Feb 25. PMID 33629188